CLINICAL TRIAL: NCT00266474
Title: Prevalence of Chronic Rhinosinusitis in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, PD Dr. Jochen G. Mainz, Head of CF Center, Pediatric Pulmonology, University of Jena
Other Study IDs: CF_Sinusitis_QS
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Cystic Fibrosis; Sinusitis
Keywords: Cystic Fibrosis with Chronic Rhinosinusitis
MeSH Terms: conditions — Cystic Fibrosis; Sinusitis | interventions — Health Records, Personal; Rhinomanometry; Nasal Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Pseudomonas aeruginosa and Staphylococcus aureus cultures (SNPS)

GROUPS / COHORTS (1):
- Cross sectional CF study: Multicentric study, including 187 CF patients of all age groupr in 5 CF centres.
  Interventions: Other: Assessment of upper and lower airway colonization, sinonasal symptoms, history, rhinoscopy and rhinomanometry.

INTERVENTIONS:
Other: Assessment of upper and lower airway colonization, sinonasal symptoms, history, rhinoscopy and rhinomanometry.
  Other Names: nasal lavage and induced sputum

SUMMARY:
Aim of the study is to detect the prevalence of chronic rhinosinusitis and the colonisation with Pseudomonas aerug. in the upper airways in patients with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of cystic fibrosis

Exclusion Criteria:

* current systemic therapy against Pseudomonas aeruginosa

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2005-12; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Pathogen colonization in upper and lower airways | 3yrs
Sinonasal symptoms (SNOT-20) | 3 yrs
rhinomanometry and rhinoscopy | 3yrs

CONTACTS AND LOCATIONS:
Overall Officials: Jochen G. Mainz, M.D., Study Chair — University of Jena
Locations (1):
- Friedrich-Schiller-Universität, Jena, Thuringia, Germany

REFERENCES:
- [Background] Mainz JG, Naehrlich L, Schien M, Kading M, Schiller I, Mayr S, Schneider G, Wiedemann B, Wiehlmann L, Cramer N, Pfister W, Kahl BC, Beck JF, Tummler B. Concordant genotype of upper and lower airways P aeruginosa and S aureus isolates in cystic fibrosis. Thorax. 2009 Jun;64(6):535-40. doi: 10.1136/thx.2008.104711. Epub 2009 Mar 11. PMID 19282318